CLINICAL TRIAL: NCT05760391
Title: A Trial of Combination and Timing of Immunotherapy With Radiotherapy in Patients With Advanced Esophageal Squamous Cell Carcinoma.
Brief Title: A Study of IO Plus Radiotherapy in Patients With Advanced ESCC.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai 19
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients will be treated with anti-PD-1 Immune Checkpoint Inhibitors combined with chemotherapy used as 1st line treatment for metastatic ESCC.Radiotherapy will be conducted after four cycles of IO plus chemotherapy or started simultaneously.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — IMRT or SABR for patients with ESCC.

SUMMARY:
This study is a single-arm, prospective, phase II trial for patients with metastatic esophageal squamous cell carcinoma (ESCC) who received immunotherapy plus chemotherapy as the first-line treatment. The aim of the study is to determine if intervening with combined local therapy and immunotherapy and chemotherapy in patients with ESCC led to significant improvements in survival and disease control compared with historical data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80, had an Eastern Cooperative Oncology Group performance status score of 0-1;
2. Patients had unresectable or recurrent esophageal squamous cell carcinoma that precluded esophagectomy or definitive chemoradiation, or distant metastatic disease;
3. Patients had received no previous systemic therapy (patients who had progressed ≥6 months after [neo]adjuvant therapy or definitive chemoradiation were eligible);
4. Patients accepted at least one cycle of anti-PD-1 immunotherapy combined chemotherapy as 1st line treatment.
5. All lesions of current diagnosis did not receive local treatment such as radiotherapy, surgery, radiofrequency ablation before enrollment.
6. The measurable lesion was determined by the investigator based on the RECIST 1.1 assessment. A lesion located in a previous radiotherapy area can be considered a target lesion if it is confirmed to progress and is considered to be measurable according to RECIST 1.1.
7. Estimated survival time >12 weeks.
8. The function of vital organs meets the following requirements:

   Neutrophil absolute count (ANC) ≥ 1.5 × 10^9 / L platelets ≥ 100 × 10^9 / L; Hemoglobin ≥ 9g / dL; serum albumin ≥ 2.8g / dL; Total bilirubin ≤ 1.5 × ULN, ALT, AST and / or AKP ≤ 2.5 × ULN; if there is liver metastasis, ALT and / or AST ≤ 5 × ULN; if there is liver metastasis or bone metastasis AKP ≤ 5 × ULN; serum creatinine ≤ 1.5 × ULN or creatinine clearance > 60 mL / min; For patients with pulmonary lesions or previous lung irradiation who are known or suspected to have impaired lung function, the forced expiratory volume (FEV1) for 1 second of lung function must be above 1L.
9. Female subjects of childbearing age must have a negative urine or serum pregnancy test within 72 hours prior to randomization. Subjects agreed to adequate contraception during the trial.
10. The patient is voluntarily enrolled and obtained the informed consent form signed by the patient or his legal representative.

Exclusion Criteria:

1. Patients who are prior exposure to immune-mediated therapy.
2. Patients participated in any investigational drug study within 4 weeks preceding the start of treatment.
3. The toxicity of previous anti-tumor treatment has not recovered to ≤ National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 level 1 (except for hair loss) or the level specified by the inclusion/exclusion criteria.
4. Patients with uncontrolled brain metastases, or vertebral body metastasis with spinal cord compression symptoms.
5. Patients with uncontrolled pleural, pericardial or pelvic effusion that requires repeated drainage.
6. Patients with history of immunodeficiency, or severe medical diseases that are not well controlled, which may have effect on the treatment of this study.
7. Any other malignant tumor was diagnosed within 5 years prior to or after the diagnosis of ESCC, except for malignant tumors with a low risk of metastasis and death (5-year survival rate >90%), such as well-treated basal cells or squamous cell skin cancer or cervical cancer in situ.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
OS from start of 1st line treatment in metastatic ESCC | 2 years
  Median OS and OS rate at 12 months and 24 months will be analysed based on Kaplan-Meier method and presented along with its 95% confidence interval.

SECONDARY OUTCOMES:
PFS from start of 1st line treatment in metastatic ESCC | 18 months
  Median PFS and PFS rate at 6 months, 12months and 18 months will be analysed based on Kaplan-Meier method and presented along with its 95% confidence interval.
Disease control rate | Evaluation at the end of radiotherapy and after every 2 months of systemic therapy.
  the ratio of patients with the best therapeutic evaluation is CR, PR and SD

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai cancer center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No